CLINICAL TRIAL: NCT01854593
Title: Prospective Randomized Controlled Study of Intravitreal Injection of 0.16 mg Bevacizumab One Day Before Surgery for Proliferative Diabetic Retinopathy
Brief Title: Prospective Randomized Controlled Study of Intravitreal Injection of Bevacizumab for Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nihon University (Other)
Responsible Party: Principal Investigator, Ayumu Manabe, Ayumu Manabe, Nihon University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCT-NAPN-23170
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-06

CONDITIONS: Proliferative Diabetic Retinopathy; Diabetic Traction Retinal Detachment; Vitreous Hemorrhage
MeSH Terms: conditions — Vitreous Hemorrhage | interventions — Bevacizumab; Vitrectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab injection and vitrectomy (Active Comparator): 0.16 mg/0.05 ml bevacizumab intravitreal injection one day before vitrectomy.
  Interventions: Drug: Bevacizumab; Procedure: Vitrectomy
- Sham injection and vitrectomy (Sham Comparator): Sham injection one day before vitrectomy.
  Interventions: Procedure: Vitrectomy; Device: Sham injection

INTERVENTIONS:
Drug: Bevacizumab — 0.16 mg/0.05 ml bevacizumab (single injection on 1 day before operation)
  Other Names: Avastin
  Arms: Bevacizumab injection and vitrectomy
Procedure: Vitrectomy — vitrectomy of 25 gauge system.
Device: Sham injection — Sham injection one day before vitrectomy
  Arms: Sham injection and vitrectomy

SUMMARY:
We hypothesized that to reduce the adverse effects of intravitreal bevacizumab on ocular tissue and whole body, intravitreal injection of a low concentration of bevacizumab and conducting vitrectomy shortly after the injection is useful. In the present prospective, double-masked, randomized, controlled study, we aimed to verify the usefulness of intravitreal injection of 0.16 mg/0.05 ml bevacizumab one day before conducting vitrectomy for PDR.

DETAILED DESCRIPTION:
Early postoperative hemorrhage in proliferative diabetic retinopathy (PDR) patients is a major complication. Intravitreal injection of anti-vascular endothelial growth factor (VEGF) has reported to reduce vitreous hemorrhage. Recently, numerous reports have shown the efficacy of reducing neovascularization activity before vitrectomy by preoperative intravitreal injection of anti-VEGF agents. When intravitreal bevacizumab (IVB) injection is used as an adjunct therapy, a shortterm effect is needed. Because it is reported some adverse events caused by bevacizumab injection. Hattori et al reported intravitreal injection of 0.16 mg/0.05 ml bevacizumab in PDR patients marked blockage of intravitreal VEGF concentrations in the pilot study. The purpose of this study is to evaluate low dose of intravitreal bevacizumab as a preoperative adjunct therapy reduce the postoperative vitreous hemorrhage. This study involves PDR patients who underwent vitrectomy between May 2012 and August 2013 at Surugadai Hospital of Nihon University. The risks to participants are accompanied by the intravitreal injection of bevacizumab (especially the possibility of endophthalmitis and thromboembolic events).

Between June 2012 and August 2013, one investigator (AM) randomized PDR patients with an indication for primary 25-gauge vitrectomy into a sham group and an IVB group. One day after injection, three surgeons except AM conducted the surgeries. Vitreous samples were collected at the start of surgery, and intraoperative and postoperative complications were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Proliferative Diabetic Retinopathy (PDR)
* Indicated for vitrectomy

Exclusion Criteria:

* History of intraocular surgery, intravitreal injection of drugs or sub-Tenon injection of steroids or retinal photocoagulation within 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayumu Manabe, Study Chair
Locations (1):
- Surugadai Nihon University Hospital, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab and Vitrectomy: 0.16mg/0.05ml bevacizumab intravitreal injection one day before surgery and vitrectomy.
  Bevacizumab: 0.16mg/0.05ml bevacizumab (single injection on 1 day before operation)
  Vitrectomy: vitrectomy of 25 gauge system.
- Sham Injection and Vitrectomy: Sham injection one day before operation and vitrectomy.
  Sham injection: Sham injection one day before vitrectomy
  Vitrectomy: vitrectomy of 25 gauge system.
Period: Overall Study
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy
Started | 34 | 35
Completed | 32 | 34
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bevacizumab and Vitrectomy: 0.16 mg/0.05 ml bevacizumab intravitreal injection one day before surgery and vitrectomy.
  * Bevacizumab: 0.16 mg/0.05 ml bevacizumab (single injection on 1 day before operation)
  * Vitrectomy: vitrectomy of 25 gauge system.
- Sham Injection and Vitrectomy: Sham injection one day before operation and vitrectomy.
  * Sham injection: Sham injection one day before vitrectomy
  * Vitrectomy: vitrectomy of 25 gauge system.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.8) | 59.2 (12.9) | 59.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 22 | 32 | 54
Preoperative best corrected visual acuity [Log Mean (Standard Deviation); unit: LogMAR] — Preoperative best corrected visual acuity
  LogMAR | 1.09 (0.60) | 1.14 (0.58) | 1.11 (0.59)
Intra Ocular Pressure [Mean (Standard Deviation); unit: mm Hg] | 15.3 (2.69) | 14.6 (3.42) | 15.0 (3.11)
Hypertension [Number; unit: participants]
  Yes | 14 | 16 | 30
  No | 18 | 18 | 36
Hyperlipidemia [Number; unit: participants]
  Yes | 5 | 7 | 12
  No | 27 | 27 | 54
HbA1c [Mean (Standard Deviation); unit: %] | 8.0 (1.7) | 7.6 (2.0) | 7.8 (1.6)
Use of anticoagulants [Number; unit: participants]
  Yes | 7 | 8 | 15
  No | 25 | 26 | 51
Lens status [Number; unit: participants]
  phakic | 28 | 31 | 59
  pseudophakic | 4 | 3 | 7
Persistent vitreous hemorrhage [Number; unit: participants] | 29 | 30 | 59
Previous panretinal photocoagulation [Number; unit: participants]
  None | 9 | 11 | 20
  Incomplete | 23 | 23 | 46
preoperative Iris neovascularization or neovascular glaucoma [Number; unit: participants] | 2 | 2 | 4

OUTCOME MEASURES:

1. Secondary Outcome: Intra Operative Hemorrhage
Description: Calculate the number of coagulators for the intra operative hemorrhage.
Time Frame: End of the surgery.
Measure: Mean (Standard Deviation); unit: coagulators
Groups:
- Sham Injection and Vitrectomy: Sham injection one day before operation and vitrectomy.
  Vitrectomy: vitrectomy of 25 gauge system.
  Sham injection: Sham injection one day before vitrectomy
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
coagulators | 0.63 (1.0) | 1.3 (1.4)
Statistical Analysis 1: Comparison: Bevacizumab and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.025, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Postoperative Vitreous Hemorrhage.
Description: Postoperative vitreous hemorrhage that is permitted within 4 weeks after surgery.
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
participants | 3 | 13
Statistical Analysis 1: Comparison: Bevacizumab and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.006, Chi-squared

3. Primary Outcome: Reoperation
Description: Vitreoretinal reoperation due to recurrent vitreous hemorrhage.
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
participants | 1 | 7
Statistical Analysis 1: Comparison: Bevacizumab and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.033, Fisher Exact

4. Secondary Outcome: Vascular Endothelial Growth Factor Concentration in Vitreous
Description: Vascular endothelial growth factor concentration in vitreous at the start of vitrectomy.
Time Frame: Start of surgery.
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
μg/ml | 25.0 (13.6) | 1315 (1153)
Statistical Analysis 1: Comparison: Bevacizumab and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Endolaser Photocoagulation
Description: Number of intraoperative endolaser photocoagulation.
Time Frame: End of surgery.
Measure: Mean (Standard Deviation); unit: photocoagulation
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
photocoagulation | 1260 (686) | 1335 (663)
Statistical Analysis 1: Comparison: Bevacizumab and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.667, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Iatrogenic Retinal Tears
Description: The number of participants who had intraoperative iatrogenic retinal tears.
Time Frame: End of surgery.
Measure: Number; unit: participants
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
participants | 5 | 5
Statistical Analysis 1: Comparison: Bevacizumab and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.593, Fisher Exact

7. Secondary Outcome: Surgical Time
Time Frame: End of surgery.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
minutes | 49 (20) | 56 (27)
Statistical Analysis 1: Comparison: Bevacizumab and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.298, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Postoperative Best Corrected Visual Acuity
Description: Best corrected visual acuity was measured using the Landolt ring chart, and the result was converted to logMAR notation for analysis.
  The minimum of the scale is 2.0 and the maximum of the scale is -0.3. The higher values represent a worse outcome.
Time Frame: 1 mouth after surgery.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
LogMAR | 0.46 (0.54) | 0.43 (0.48)
Statistical Analysis 1: Comparison: Bevacizumab and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.929, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Best Corrected Visual Acuity Change
Description: Best corrected visual acuity change was calculated by postoperative logMAR visual acuity minus preoperative logMAR visual acuity.
  The higher values represent a worse outcome.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
LogMAR | -0.63 (0.61) | -0.73 (0.80)
Statistical Analysis 1: Comparison: Bevacizumab and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.445, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Postoperative Neovascular Glaucoma
Description: The number of participants with progressive or persistent neovascular glaucoma after surgery.
Time Frame: Within 1 month after the surgery.
Measure: Number; unit: participants
Groups:
- Bevacizumab Injection and Vitrectomy: 0.16mg/0.05ml bevacizumab intravitreal injection one day before surgery and vitrectomy.
  Bevacizumab: 0.16mg/0.05ml bevacizumab (single injection on 1 day before operation)
  Vitrectomy: vitrectomy of 25 gauge system.
Arm/Group | Bevacizumab Injection and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
participants | 0 | 3
Statistical Analysis 1: Comparison: Bevacizumab Injection and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.131, Chi-squared

11. Secondary Outcome: Elevated Intraocular Pressure
Description: The number of participants with elevated intraocular pressure after surgery.
Time Frame: Within 1 month after the surgery.
Measure: Number; unit: participants
Arm/Group | Bevacizumab Injection and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
participants | 2 | 6
Statistical Analysis 1: Comparison: Bevacizumab Injection and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.149, Fisher Exact

12. Secondary Outcome: Gas Tamponade
Description: The number of participants with gas tamponade at the end of the surgery.
Time Frame: End of surgery.
Measure: Number; unit: participants
Arm/Group | Bevacizumab Injection and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
participants | 23 | 24
Statistical Analysis 1: Comparison: Bevacizumab Injection and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.670, Fisher Exact

13. Secondary Outcome: Silicon Oil Tamponade
Description: The number of participants with silicon oil tamponade at the end of the surgery.
Time Frame: End of surgery.
Measure: Number; unit: participants
Arm/Group | Bevacizumab Injection and Vitrectomy | Sham Injection and Vitrectomy
Number analyzed (Participants) | 32 | 34
participants | 4 | 6
Statistical Analysis 1: Comparison: Bevacizumab Injection and Vitrectomy vs Sham Injection and Vitrectomy; Test type: Superiority or Other; p = 0.378, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 month
Description: 1 month after vitrectomy.
Arm/Group | Bevacizumab and Vitrectomy | Sham Injection and Vitrectomy
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34
Other Adverse Events (participants affected / at risk) | 0/32 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes